CLINICAL TRIAL: NCT02353910
Title: VTE Incidence and Risk Factors in Patients With Severe Sepsis and Septic Shock
Brief Title: VTE Incidence in Severe Sepsis and Septic Shock
Status: Completed | Type: Observational
Sponsor: University of Utah (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Matthew Rondina, MD, Associate Professor, University of Utah
Other Study IDs: 1001
Record Dates: First submitted 2015-01-23; First posted 2015-02-03 (Estimated); Last update posted 2015-02-03 (Estimated); Status verified 2015-01

CONDITIONS: Severe Sepsis With Septic Shock
MeSH Terms: interventions — High-Energy Shock Waves

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Procedure: Ultrasound

SUMMARY:
Prospective studies on the incidence of VTE during severe sepsis and septic shock remain absent, hindering efficacy assessments regarding current VTE prevention strategies in septic patients. The investigators will prospectively study consecutively enrolled ICU patients with severe sepsis and septic shock admitted at three hospitals. All patients will provide informed consent and the study will be IRB approved. VTE thromboprophylaxis, provided per standard of care and according to the patients' primary team, will be recorded for all patients. Patients will undergo bilateral lower (and upper, if a central venous catheter [CVC] was present) comprehensive compression ultrasonography (CUS) and will be followed for symptomatic deep vein thrombosis (DVT) and pulmonary embolism (PE) prior to discharge. The investigators will perform multivariate regression analyses to identify predictors of VTE.

ELIGIBILITY:
Inclusion Criteria:

* ICU patients with severe sepsis and septic shock

Exclusion Criteria:

* Admission diagnosis of acute VTE,
* age < 13 years,
* pregnancy,
* severe chronic respiratory disease,
* severe chronic liver disease (Child-Pugh Score of 11-15),
* moribund patients not expected to survive 24 hours, and
* acute myocardial infarction within 30 days.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: We prospectively studied 113 consecutively enrolled ICU patients with severe sepsis and septic shock admitted at three hospitals. All patients provided informed consent and this study was IRB approved. VTE thromboprophylaxis was recorded for all patients. Patients underwent bilateral lower (and upper, if a central venous catheter [CVC] was present) comprehensive compression ultrasonography (CUS) and were followed for symptomatic deep vein thrombosis (DVT) and pulmonary embolism (PE) prior to discharge. We performed multivariate regression analyses to identify predictors of VTE
Sampling Method: Probability Sample
Enrollment: 113 (Actual)
Dates: Start 2009-07; Primary Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Incidence of VTE | 28 days

REFERENCES:
- [Derived] Kaplan D, Casper TC, Elliott CG, Men S, Pendleton RC, Kraiss LW, Weyrich AS, Grissom CK, Zimmerman GA, Rondina MT. VTE Incidence and Risk Factors in Patients With Severe Sepsis and Septic Shock. Chest. 2015 Nov;148(5):1224-1230. doi: 10.1378/chest.15-0287. PMID 26111103